CLINICAL TRIAL: NCT04658966
Title: Validation of the French Translation of a Self-questionnaire Looking for a History of Pre-eclampsia of More Than 5 Years in Women Who Have Already Had a Pregnancy of More Than 6 Months With Childbirth at Brest University Hospital.
Brief Title: Validation of the French Translation of a Self-questionnaire Looking for a History of Pre-eclampsia.
Acronym: PRERETRO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PRERETRO ( 29BRC20.0133)
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Preeclampsia
Keywords: questionnaire
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: Women with a history of pre-eclampsia
  Interventions: Other: administration of a self-questionnaire
- controls: Women with no history of hypertensive disorder during pregnancy
  Interventions: Other: administration of a self-questionnaire

INTERVENTIONS:
Other: administration of a self-questionnaire — Women will have to fill in an online self questionnaire on pre-eclampsia

SUMMARY:
PRERETRO is a study for validation of the French translation of a self-questionnaire looking for a history of pre-eclampsia of more than 5 years in women who have already had a pregnancy of more than 6 months with childbirth at Brest University Hospital.

DETAILED DESCRIPTION:
This study will help to evaluate the specificity and sensitivity of the French translation of a self-questionnaire looking for a history of pre-eclampsia in women who gave birth at Brest University Hospital before year 2015.

First, women with pre-eclampsia (cases) and women with no hypertensive disorders (controls) during pregnancy were identified with the Medical Registry Database (MRD) of Brest University maternity ward.

All pre-eclampsia diagnoses were reviewed by 2 experts in order to confirm the accuracy of the diagnosis.

250 cases and 250 controls were finally selected after consultation of their medical file and were pre-included in the study.

Then, the 500 women will be contacted by phone or e-mail in order to inform them about the study and to offer them the possibility to participate in the study.

The women who will agree to participate in the study will fill in an online self-questionnaire on pre-eclampsia.

Their responses will then be compared to the diagnosis retained after consultation of their medical file.

Sensitivity and specificity of the questionnaire will then be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women who gave birth after a pregnancy of more than 6 months at Brest University Hospital between January 2002 and December 2014
* For the cases: with a pre-eclampsia diagnosis during pregnancy
* For the controls: with no history of hypertensive disorder during pregnancy

Exclusion Criteria:

* Women Under legal protection
* Women unable to read French
* Medical interruption of pregnancy
* Pregnancy with a delivery before 6 months
* Women who refused to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who gave birth after a pregnancy of more than 6 months at Brest University Hospital between January 2002 and December 2014
Study Population: Cases will be women with a history of pre-eclampsia before 2015 and controls will be women with no history of hypertensive disorder during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Evaluate diagnostic sensitivity and specificity of the self questionnaire | Inclusion ( Day 0)
  Presence or not of a history pre-eclampsia according to responses to the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the end study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Result] Societe francaise d'anesthesie et de reanimation (Sfar); College national des gynecologues et obstetriciens francais (CNGOF); Societe francaise de medecine perinatale (SFMP); Societe francaise de neonatalogie (SFNN). [Multidisciplinary management of severe pre-eclampsia (PE). Experts' guidelines 2008. Societe francaise d'anesthesie et de reanimation. College national des gynecologues et obstetriciens francais. Societe francaise de medecine perinatale. Societe francaise de neonatalogie]. Ann Fr Anesth Reanim. 2009 Mar;28(3):275-81. doi: 10.1016/j.annfar.2009.02.015. Epub 2009 Mar 24. No abstract available. French. PMID 19321292
- [Result] Saucedo M, Deneux-Tharaux C, Bouvier-Colle MH; Le Comite national d'experts sur la mortalite maternelle. [Maternal mortality in France, 2007-2009]. J Gynecol Obstet Biol Reprod (Paris). 2013 Nov;42(7):613-27. doi: 10.1016/j.jgyn.2013.06.011. Epub 2013 Sep 13. French. PMID 24035736
- [Result] Bellamy L, Casas JP, Hingorani AD, Williams DJ. Pre-eclampsia and risk of cardiovascular disease and cancer in later life: systematic review and meta-analysis. BMJ. 2007 Nov 10;335(7627):974. doi: 10.1136/bmj.39335.385301.BE. Epub 2007 Nov 1. PMID 17975258
- [Result] van Wyk L, van der Marel J, Schuerwegh AJ, Schouffoer AA, Voskuyl AE, Huizinga TW, Bianchi DW, Scherjon SA. Increased incidence of pregnancy complications in women who later develop scleroderma: a case control study. Arthritis Res Ther. 2011;13(6):R183. doi: 10.1186/ar3510. Epub 2011 Nov 4. PMID 22053948
- [Result] Kamper-Jorgensen M, Gammill HS, Nelson JL. Preeclampsia and scleroderma: a prospective nationwide analysis. Acta Obstet Gynecol Scand. 2018 May;97(5):587-590. doi: 10.1111/aogs.13296. Epub 2018 Feb 8. PMID 29344946
- [Result] Diehl CL, Brost BC, Hogan MC, Elesber AA, Offord KP, Turner ST, Garovic VD. Preeclampsia as a risk factor for cardiovascular disease later in life: validation of a preeclampsia questionnaire. Am J Obstet Gynecol. 2008 May;198(5):e11-3. doi: 10.1016/j.ajog.2007.09.038. Epub 2008 Feb 1. PMID 18241822